CLINICAL TRIAL: NCT06296420
Title: Dysphagia After Thyroidectomy
Acronym: DYSPHATHYR
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 24C304
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Goiter; Thyroid Disease
Keywords: Nodular goiter; Thyroidectomy; Dysphagia; Psychometrics; Rasch analysis
MeSH Terms: conditions — Goiter; Thyroid Diseases; Goiter, Nodular; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to develop a questionnaire for measuring swallowing and throat discomfort symptoms in patients with goiter or thyroidectomy, which complies with the model of Rasch and which satisfies the fundamental measurement axioms (e.g., unidimensionality, linearity, generalizability). Developing a scale with such characteristics would provide clinicians and researchers with a reliable tool for assessing the impact of goiter and for measuring the outcomes after surgery.

Also, the study will assess the psychological impact of goiter and thyroidectomy, as well as the characteristics of the surgical scar after thyroidectomy.

The questionnaire will be developed in the first phase of the study. Items and response categories will be identified through interviews performed with patients affected by goiter or after thyroidectomy.

In the following phases of the study, the questionnaire will be administered to patients before and after thyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of goiter or thyroidectomy.

Exclusion Criteria:

* Diagnosis of other neurological disorders or disorders involving the aerodigestive tract that could cause swallowing disorders.
* Previous surgery of the neck or involving the aerodigestive tract.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the first phase, the study will recruit patients with diagnosis of goiter who are candidates to thyroidectomy and patients who have undergone thyroidectomy. Patients will be interviewed by the researchers. The interviews will face the symptoms of goiter or thyroidectomy, dealing (not exclusively) with throat and swallowing symptoms. The interviews will be recorded and analysed. The content of the interviews will be used to develop the items and the response categories of the questionnaire.
  In the second phase, the study will recruit patients who are candidates for thyroidectomy. The questionnaire (and the other outcome measures of the study) will be administered to the patients before and after surgery. All patients who are candidates for thyroidectomy at the Istituto Auxologico Italiano in Milan, Italy, will be recruited (if they comply with inclusion and exclusion criteria and if they provide consent). General, clinical and surgical data will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure will be the questionnaire which will be developed in the first phase of the study itself. | In the week before surgery, three months after surgery, and six months after surgery.
  The questionnaire will be administered to the recruited patients three times: in the week before surgery, three months after surgery, and six months after surgery.

SECONDARY OUTCOMES:
Patient and Observer Scar Assessment Scale (POSAS) 2.0. | The POSAS 2.0 will be administered 10 days after surgery and 2 months after surgery.
  The Patient and Observer Scar Assessment Scale (POSAS) 2.0. is an assessment scale that measures the quality of the scar from the perspectives of the patient and the clinician. It is made of two separate subscales, i.e., the Observer Scar Assessment Scale and the Patient Scar Assessment Scale. The Observer Scar Assessment Scale is made of 6 items, each scored 1 to 10 (total score 6 to 60, with higher scores indicating worse scar quality). The Patient Scar Assessment Scale is made of 7 items, each scored 1 to 10, divided in three subsets (total score 7 to 70, with higher scores indicating worse scar quality).
Depression Anxiety Stress Scales-21 (DASS-21). | The DASS-21 will be administered 10 days before surgery and 2 months after surgery.
  The Depression Anxiety Stress Scales-21 (DASS-21) is an assessment scale used to measure the severity of symptoms of depression, anxiety and stress. It is made of 21 items, each scored 0 to 3 (total score 0 to 63, with higher scores for greater severity of depression, anxiety and/or stress.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Scarano, MD, Principal Investigator — University of Milan, IRCCS Istituto Auxologico Italiano
Locations (1):
- IRCCS Istituto Auxologico Italiano, Milan, MI, Italy